CLINICAL TRIAL: NCT04064450
Title: MyoVasc - An Epidemiological Cohort Study to Investigate the Development and Progression of Heart Failure and the Interaction With Vascular Disease
Brief Title: MyoVasc Study on the Development and Progression of Heart Failure
Status: Active, not recruiting | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Philipp Wild, MD, MSc, Univ.-Prof. Dr. Philipp S. Wild, MD, MSc, Johannes Gutenberg University Mainz
Other Study IDs: 837.319.12 (8420-F)
Record Dates: First submitted 2019-08-09; First posted 2019-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Heart Failure
Keywords: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Heart Failure: Individuals with asymptomatic or symptomatic heart failure
- Population Controls: Individuals free of heart failure and echocardiographic cardiac dysfunction

SUMMARY:
The MyoVasc - Study is an observational, prospective cohort study. The study is investigating the development and progression of the heart failure syndrome, phenotypes of the heterogeneous syndrome, and the interactions of phenotypes with the vasculature regarding their impact for the course of heart failure.

DETAILED DESCRIPTION:
"MyoVasc" is an observational cohort study investigating the development and progression of heart failure (HF). The primary objective of the study is: i, to advance the understanding of pathomechanisms of the heterogenous syndrome in the full range of clinical presentation, ii, to evaluate current clinical phenotypes of HF, and iii, to identify and describe homogenous subgroups with regard to disease development using a systems-oriented approach. A special focus is put on the investigation of heart failure with preserved ejection fraction in contrast to the more investigated and established phenotype with reduced ejection fraction. Further aspects comprise inter alia the relevance of metabolic dysregulation, inflammation and coagulation for the course of the disease.

The primary endpoint of the study is the combined outcome "worsening of heart failure" defined as transition from asymptomatic to symptomatic heart failure, hospitalization due to heart failure, or cardiac death. Secondary endpoints are the components of the primary endpoint, myocardial infarction, stroke, hospitalization due to cardiovascular disease, venous thromboembolism, atrial fibrillation, and all-cause death. Disease progression is monitored by a large panel of biomarkers for structure and function of cardiac and vascular systems and related organs.

Individuals aged 35- to 84-years with echocardiographic signs of heart failure irrespective of the clinical status are enrolled and a subsample of controls without heart failure. Individuals were recruited from health institutions and a population sample from the registration office. The study sample comprises approx. 3,200 individuals, of which N~2,700 individuals have heart failure and N~500 individuals are controls. Study participants receive a highly standardized 5-hour baseline examination in the study center with examinations of the cardiovascular system (e.g. anthropometrics, 2D- and 3D-echocardiography, carotid sonography, vascular function, ankle-brachial index, body plethysmography, capacity exercise testing, blood pressure measurements (resting, ABPM), ECG (12-lead, holter), computer-assisted personal interview, and venous blood withdrawal for bio banking). Annual follow-up examinations are performed via computer-assisted telephone interviews tracking comprehensively the participants´ health status, assessing current medication and recording clinical events. Every two years, the participant is invited again to the MyoVasc Study Center for the conduct of sequential follow-up investigations, which are identical to the initial examination.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic heart failure or symptomatic heart failure
* Written consent
* Sufficient knowledge of the German language, in order to understand study documents and computer assisted interview without any translation

Exclusion Criteria:

* Individuals who are not able to visit the study center due to psychological or physical impairment
* STEMI within the last 4 months, NSTEMI within the last 3 months
* Acute decompensated heart failure
* Surgery, especially coronary artery bypass grafting within the last 3 months
* Acute disease, especially acute infectious disease, endocarditis, myocarditis or pericarditis

Ages: 35 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with asymptomatic and symptomatic heart failure and Population Controls
Sampling Method: Non-Probability Sample
Enrollment: 3289 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Worsening of Heart Failure | Assessment in annual follow-up contacts over a period of 10 years
  The primary outcome "worsening of heart failure" differs between groups:
  * Population Controls: i.e. composite of cardiac death and incident heart failure (i.e. incident asymptomatic or symptomatic heart failure)
  * Individuals with asymptomatic heart failure: i.e. composite of cardiac death and transition from asymptomatic to symptomatic heart failure
  * Individuals with symptomatic heart failure: i.e. composite of cardiac death and hospitalization due to worsening of heart failure

SECONDARY OUTCOMES:
Incidence of Cardiac death | Assessment in annual follow-up contacts over a period of 10 years
  Cardiac death
Incidence of Hospitalization due to heart failure | Assessment in annual follow-up contacts over a period of 10 years
  Hospitalization due to heart failure
Incidence of transition from asymptomatic to symptomatic heart failure | Assessment in annual follow-up contacts over a period of 10 years
  Transition from asymptomatic to symptomatic heart failure
Incidence of heart failure (i.e. incident asymptomatic or symptomatic heart failure) in controls | Assessment in annual follow-up contacts over a period of 10 years
  Incident heart failure (i.e. incident asymptomatic or symptomatic heart failure) in controls
Incidence of death | Follow-up of vital status for 10 years
  Death
Incidence of hospitalization | Assessment in annual follow-up contacts over a period of 10 years
  Hospitalization
Incidence of myocardial infarction | Assessment in annual follow-up contacts over a period of 10 years
  Myocardial infarction
Incidence of stroke or transient ischemic attack | Assessment in annual follow-up contacts over a period of 10 years
  Stroke or transient ischemic attack
Incidence of cardiac arrhythmia | Continuous assessment throughout the follow-up of the study
  Cardiac arrhythmia
Incidence of atrial fibrillation | Assessment in annual follow-up contacts over a period of 10 years
  Atrial fibrillation
Incidence of angina pectoris | Assessment in annual follow-up contacts over a period of 10 years
  Angina pectoris
Incidence of deep vein thrombosis | Assessment in annual follow-up contacts over a period of 10 years
  Deep vein thrombosis
Incidence of pulmonary embolism | Assessment in annual follow-up contacts over a period of 10 years
  Pulmonary embolism
Incidence of arterial hypertension | Assessment in annual follow-up contacts over a period of 10 years
  Arterial hypertension
Incidence of peripheral artery disease | Assessment in annual follow-up contacts over a period of 10 years
  Peripheral artery disease
Worsening of exercise capacity as assessed via peak oxygen uptake | Assessment in biannual follow-up contacts in a dedicated study center after 2, 4, 6, 8 and 10 years
  Assessment of peak oxygen uptake via cardiopulmonary exercise testing under consideration of the circulatory (blood pressure, heart rate, electrocardiogram) and respiratory response (ventilatory anaerobic threshold and reserve) by a trained physician
Worsening of systolic cardiac function assessed by ventricular ejection fraction | Assessment in biannual follow-up contacts in a dedicated study center after 2, 4, 6, 8 and 10 years
  Assessed via 2D/3D transthoracic cardiac echocardiography by a trained physician
Incidence of revascularization | Assessment in annual follow-up contacts over a period of 10 years
  Revascularization
Worsening of diastolic cardiac function assessed by mitral inflow signal and tissue doppler of the heart | Assessment in biannual follow-up contacts in a dedicated study center after 2, 4, 6 and 8 years
  Assessed via 2D/3D transthoracic cardiac echocardiography by a trained physician
Worsening of cardiac strain assessed by speckle-tracking of the heart | Assessment in biannual follow-up contacts in a dedicated study center after 2, 4, 6, 8 and 10 years
  Assessed via 2D/3D transthoracic cardiac echocardiography by a trained physician
Worsening of renal function as assessed by glomerular filtration rate | Assessment in biannual follow-up contacts in a dedicated study center after 2, 4, 6, 8 and 10 years
  Worsening of renal function as assessed by estimated glomerular Filtration rate (eGFR) as humoral biomarker of renal function
Worsening of pulmonary function as assessed by FEV1 | Assessment in biannual follow-up contacts in a dedicated study center after 2, 4, 6, 8 and 10 years
  Worsening of forced expiratory volume in one second (FEV1) via body plethysmography
Worsening of vascular function as assessed by FMD/FMC | Assessment in biannual follow-up contacts in a dedicated study center after 2, 4, 6, 8 and 10 years
  Worsening of flow-mediated dilatation (FMD) and constriction (FMC) of the radial artery

CONTACTS AND LOCATIONS:
Overall Officials: Philipp S Wild, MD, MSc, Principal Investigator — University Medical Center of the Johannes Gutenberg University Mainz
Locations (1):
- University Medical Center of the Johannes Gutenberg-University Mainz, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trobs SO, Prochaska JH, Schwuchow-Thonke S, Schulz A, Muller F, Heidorn MW, Gobel S, Diestelmeier S, Lerma Monteverde J, Lackner KJ, Gori T, Munzel T, Wild PS. Association of Global Longitudinal Strain With Clinical Status and Mortality in Patients With Chronic Heart Failure. JAMA Cardiol. 2021 Apr 1;6(4):448-456. doi: 10.1001/jamacardio.2020.7184. PMID 33533883
- [Background] Dahlen B, Schulz A, Gobel S, Trobs SO, Schwuchow-Thonke S, Spronk HM, Prochaska JH, Arnold N, Lackner KJ, Gori T, Ten Cate H, Munzel T, Wild PS, Panova-Noeva M. The impact of platelet indices on clinical outcome in heart failure: results from the MyoVasc study. ESC Heart Fail. 2021 Aug;8(4):2991-3001. doi: 10.1002/ehf2.13390. Epub 2021 May 3. PMID 33939298
- [Background] Eggebrecht L, Prochaska JH, Trobs SO, Schwuchow-Thonke S, Gobel S, Diestelmeier S, Schulz A, Arnold N, Panova-Noeva M, Koeck T, Rapp S, Gori T, Lackner KJ, Ten Cate H, Munzel T, Wild PS. Direct oral anticoagulants and vitamin K antagonists are linked to differential profiles of cardiac function and lipid metabolism. Clin Res Cardiol. 2019 Jul;108(7):787-796. doi: 10.1007/s00392-018-1408-y. Epub 2019 Jan 2. PMID 30604046
- [Background] Prochaska JH, Arnold N, Falcke A, Kopp S, Schulz A, Buch G, Moll S, Panova-Noeva M, Junger C, Eggebrecht L, Pfeiffer N, Beutel M, Binder H, Grabbe S, Lackner KJ, Ten Cate-Hoek A, Espinola-Klein C, Munzel T, Wild PS. Chronic venous insufficiency, cardiovascular disease, and mortality: a population study. Eur Heart J. 2021 Oct 21;42(40):4157-4165. doi: 10.1093/eurheartj/ehab495. PMID 34387673
- [Background] Zeid S, Buch G, Velmeden D, Sohne J, Schulz A, Schuch A, Trobs SO, Heidorn MW, Muller F, Strauch K, Coboeken K, Lackner KJ, Gori T, Munzel T, Prochaska JH, Wild PS. Heart rate variability: reference values and role for clinical profile and mortality in individuals with heart failure. Clin Res Cardiol. 2024 Sep;113(9):1317-1330. doi: 10.1007/s00392-023-02248-7. Epub 2023 Jul 9. PMID 37422841
- [Background] Heidorn MW, Steck S, Muller F, Trobs SO, Buch G, Schulz A, Schwuchow-Thonke S, Schuch A, Strauch K, Schmidtmann I, Lackner KJ, Gori T, Munzel T, Wild PS, Prochaska JH. FEV1 Predicts Cardiac Status and Outcome in Chronic Heart Failure. Chest. 2022 Jan;161(1):179-189. doi: 10.1016/j.chest.2021.07.2176. Epub 2021 Aug 17. PMID 34416218
- [Derived] Gobel S, Prochaska JH, Trobs SO, Panova-Noeva M, Espinola-Klein C, Michal M, Lackner KJ, Gori T, Munzel T, Wild PS. Rationale, design and baseline characteristics of the MyoVasc study: A prospective cohort study investigating development and progression of heart failure. Eur J Prev Cardiol. 2021 Aug 9;28(9):1009-1018. doi: 10.1177/2047487320926438. Epub 2020 May 14. PMID 34402876